CLINICAL TRIAL: NCT06373835
Title: Efficacy, Safety and Pharmacokinetics of Ascending Dosages of Emodepside and in Comparison to Ivermectin Against Strongyloidiasis Stercoralis in Adults: Randomized Stage II Seamless Adaptive Controlled Trials
Brief Title: Efficacy and Safety of Emodepside in Adults Infected With Strongyloidiasis Stercoralis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: National Institute of Public Health, Vientiane, Laos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMODEPSIDE_LAOS
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Strongyloides Stercoralis Infection; Strongyloidiasis
MeSH Terms: conditions — Strongyloidiasis | interventions — emodepside

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Emodepside 5 mg (Experimental): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Emodepside 10 mg (Experimental): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Emodepside 15 mg (Experimental): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Emodepside 20 mg (Experimental): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Emodepside 25 mg (Experimental): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Emodepside 30 mg (Experimental): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Placebo (Placebo Comparator): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside
- Ivermectin 3 mg (Active Comparator): Treatment with ascending doses of emodepside (from 5 mg to 30 mg) or ivermectin (200 μg/kg) or placebo.
  Interventions: Drug: Emodepside

INTERVENTIONS:
Drug: Emodepside — 5 mg tablets of emodepside and matching placebo tablets, 3mg ivermectin

SUMMARY:
Efficacy, safety and pharmacokinetics of ascending dosages of emodepside and in comparison to ivermectin against Strongyloidiasis stercoralis in adults: randomized stage II seamless adaptive controlled trials

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed by the participant him/herself
* Males and females of age 18 or older
* Infected with S. stercoralis (positive by at least two Baermann assays on two different days and infection intensities of at least 0.75 LPG in the two stool samples.
* Agree to comply with the study procedures, including to be examined by a study physician at the beginning of the study and to provide three stool samples during the screening period (within a maximum of 10 days) and approximately three weeks after treatment (follow-up).
* Female participants of childbearing potential to ensure adequate contraception during the study period.

Exclusion Criteria:

* No written informed consent by individual.
* Presence of acute or uncontrolled systemic illnesses (e.g. severe anemia, clinical malaria) as assessed by a medical doctor, upon initial clinical assessment.
* Recent history of acute or severe chronic disease, as assessed by a medical doctor or reported by the participant: Type 1 and/or 2 diabetes; Psychiatric disorders; Chronic heart, liver, or renal disease
* Prior treatment with anthelmintics (eg, diethylcarbamazine [DEC], suramin, ivermectin, mebendazole or albendazole) within 4 weeks before planned study drug administration.
* Actively participating in other clinical trials during the study.
* Positive pregnancy test or breastfeeding women and planning to become pregnant within three months of study drug administration.
* Received strong CYP3A4 inducers or inhibitors as well as concomitant treatments that are relevant substrate for CYP3A4 such as clarithromycin, erythromycin and rifampicin within 4 weeks before planned study drug administration.
* Received strong P-gp inhibitors as well as concomitant treatments that are relevant substrates for P-gp such as clotrimazole and ritonavir.
* Known allergy to study drugs or any of the ingredients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2024-05-20 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2024-09-21 (Actual)

PRIMARY OUTCOMES:
Cure rate (CR) of emodepside against Strongyloides stercoralis | In the week between 14 and 21 days post-treatment
  The CR will be calculated as the proportion of Strongyloides stercoralis larvae-positive participants at baseline who become larvae-negative after treatment.

SECONDARY OUTCOMES:
Safety and tolerability of the dose-dependent emodepside treatment regimes, and compared with ivermectin. | Actively evaluated at 3 hours, 24 hours, 72 hours, and 14 days post-treatment
  AEs will be evaluated descriptively as the difference of proportion reported AEs before and after treatment.
Geometric Mean Larvae Reduction Rate (LRR) of emodepside against Strongyloides stercoralis. | In the week between 14 and 21 days post-treatment
  The LRRs will be calculated based on the geometric mean
Exposure response of emodepside in adults | Actively collected at 0 hours, 0.5 hours, 2.5 hours, 5 hours, 24 hours, 72 hours, and 14 days post-treatment
  Emodepside will be quantified using a validated liquid chromatography tandem mass spectrometry (LC-MS/MS) method. Drug concentrations will be calculated by interpolation from a calibration curve with a foreseen limit of quantification of approximately 1-5 ng/ml.
Cure rate (CR) and egg reduction rate (ERR) with other soil-transmitted helminths (STH) and trematodes | In the week between 14 and 21 days post-treatment
  The CR will be calculated as the proportion of the STH or trematode positive participants at baseline who become egg-negative after treatment. The egg reduction rate (ERR) is calculated as follows: ERR = (1-(geometric mean EPG at follow-up/geometric mean EPG at baseline))*100).

CONTACTS AND LOCATIONS:
Locations (1):
- Lao Tropical and Public Health Institute, Vientiane, Laos

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Taylor L, Many S, Jeanguenat H, Hattendorf J, Sayasone S, Keiser J. Efficacy and safety of ascending doses of emodepside in comparison with ivermectin in adults infected with Strongyloides stercoralis in Laos: a phase 2a, dose-ranging, randomised, parallel-group, placebo-controlled, single-blind clinical trial. Lancet Infect Dis. 2025 Nov;25(11):1254-1264. doi: 10.1016/S1473-3099(25)00255-5. Epub 2025 Jun 25. PMID 40580974